CLINICAL TRIAL: NCT03000283
Title: Conivaptan for the Reduction of Cerebral Edema in Intracerebral Hemorrhage- A Safety and Tolerability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jesse Corry (Other)
Responsible Party: Sponsor-Investigator, Jesse Corry, Neurologist, Allina Health System
Organization: Allina Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSJC-1601
Record Dates: First submitted 2016-12-14; First posted 2016-12-22 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Cerebral Hemorrhage; Cerebral Edema; Intracerebral Hemorrhage; Stroke
Keywords: Conivaptan
MeSH Terms: conditions — Cerebral Hemorrhage; Brain Edema; Stroke | interventions — conivaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Conivaptan Treatment Group (Experimental): All seven patients in this arm will receive conivaptan as described in Interventions.
  Interventions: Drug: Conivaptan

INTERVENTIONS:
Drug: Conivaptan — Patients will receive 20mg IV of the study drug every 12 hours equaling 40mg/day over 2 days (4 doses total), in addition to the standardized ICH management targets using the PI's version of standardized ICH management targets.Usual standard of care can include sedation and analgesia as needed, elevation of the head of the bed, mannitol and/or saline as needed to reduce ICP, and temperature control with antipyretics such as acetaminophen.
  The conivaptan bolus (20mg), which is premixed with 100ml of 5% dextrose in water, is infused (peripherally) over 30 minutes, most commonly through an already placed central line.
  Other Names: Vaprisol

SUMMARY:
The goal of this study is to preliminarily determine/estimate feasibility and whether frequent and early conivaptan use, at a dose currently determined to be safe (i.e., 40mg/day), is safe and well-tolerated in patients with cerebral edema from intracerebral hemorrhage (ICH) and pressure (ICP). A further goal is to preliminarily estimate whether conivaptan at this same dose can reduce cerebral edema (CE) in these same patients. This study is also an essential first step in understanding the role of conivaptan in CE management.

Hypothesis: The frequent and early use of conivaptan at 40mg/day will be safe and well-tolerated, and also reduce cerebral edema, in patients with intracerebral hemorrhage and pressure.

DETAILED DESCRIPTION:
This is a single-center, open-label, safety and tolerability study. Based on findings in the literature from both animal research and clinical observations with ICH (intracerebral hemorrhage) associated with TBI (traumatic brain injury), this study will begin to look at the safety, tolerability, as well as potential effectiveness, of conivaptan to reduce CE (cerebral edema) in patients with non-traumatic ICH.

The seven patients in this study will receive 40mg/day of the study medication conivaptan. In this early phase study, our focus will be to assess the safety and tolerability of this medication. The available clinical data on conivaptan in the neurocritical care population suggest the potential harm is negligible. Data in TBI patients demonstrate conivaptan is safe and well tolerated using a single dose (20mg) to increase Na+ in a controlled fashion to reduce ICP. Previous work has demonstrated the safety and tolerability of conivaptan, in doses ranging from 20-80mg/day, in the neurocritical care population. Conivaptan has been demonstrated to be safe and effective in lowering ICP, and increasing serum sodium, in the neurocritical care population. Also noted have been improvements in cerebral perfusion pressure (CPP) and stable blood pressure, and a prolonged reduction in ICP. Finally, the method of intermittent bolus dosing of conivaptan is equally effective in raising and maintaining serum sodium in the neurocritical care population as continuous infusion, with potentially less risk of adverse reactions including phlebitis.

Conivaptan, a non-selective Arginine-Vasopressin (AVP) V1A/V2 antagonist that reduces aquaporin 4 production and promotes aquaresis, is approved for the treatment of euvolemic and hypervolemic hyponatremia. The exact cause of the observed reduction in ICP with conivaptan is uncertain. However, the mechanism most likely represents a combination of an acute pure aquaresis, removing free water from brain tissue, and a sustained down regulation of aquaporin 4 to abate/slow development of CE. The V2 antagonism of conivaptan promotes free water loss, and the V1 antagonism may improve cerebral blood flow (CBF) and reduce blood brain barrier permeability. Notably, serum sodium tends to correlate inversely with both ICP and CE. The early use of conivaptan could potentially be used clinically to reduce CE by these means.

It is with this in mind, the research team feels justified in pursuing this study with the hopes that the data obtained will lead to potential good and removal of harm in future patients with this devastating disease. Given the enormous costs of ICH, problems with current therapies, and variability in treatment, there is an urgent need to identify a therapy that has a better safety and effectiveness profile compared to the currently used agents. This study will use a dose (40mg/day) currently approved. Further, given that the primary purpose of the use of this medication in this study is not to correct hyponatremia, an investigational new drug (IND) application to the FDA was submitted, and the study was determined exempt.

Our central hypothesis is that through reductions in aquaporin-4 (AQP4) expression, the early use of conivaptan will reduce CE while also being safe to the patient. Our long term goal is to show that early use of conivaptan in ICH will reduce CE. If this reduction is possible, we hypothesize improved outcome and reducing the need for rescue therapies, ICU length of stay, and overall treatment cost will follow. However, more data is needed to evaluate the dosing and amount of drug. With respect to conivaptan's efficacy in correction of hyponatremia, a direct dose-response relationship exists. Further, this effect was more noted at milder degrees of hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old and < 80 years.
2. Diagnosis of primary ICH > 20 cc in volume.
3. Enrollment within 48 hours from initial symptoms.
4. Signed informed consent from the patient or obtained via their legally authorized representative (if the patient is not able to sign the informed consent themselves). The patient's decisional capacity to either provide or refuse consent will be determined using the Glasgow Coma Scale (GCS), which is being assessed at baseline and at 24 hours (+/-6hrs) after enrollment. A potential study participant with a GCS > 14 will be asked to provide their own initial study consent. A GCS ≤ 14 would indicate the need to pursue consent via legally authorized representative.

Exclusion Criteria:

1. Current need for renal replacement therapy (RRT).
2. Glomerular filtration rate (GFR) of <30 mL/minute at time of admission.
3. Participation in another study for ICH or intraventricular hemorrhage.
4. ICH related to infection, thrombolysis, subarachnoid hemorrhage, trauma or tumor.
5. Presence of HIV or active fungal infection that is known based on information in the electronic medical record (EMR).
6. Continued use of digoxin or amlodipine (as recommended by the manufacturer due to cytochrome P450 3A4 "CYP3A" inhibition).
7. Active hepatic failure as defined by aspartate aminotransferase (AST) >160 units/L and/or alanine transaminase (ALT) >180 units/L, or total bilirubin levels greater than four times normal levels (>4.8mg/dL).
8. Serum Na+> 145 mmol/L (admission labs or any time prior to recruitment/enrollment).
9. Unable to receive conivaptan based on contraindications indicated by the manufacturer.
10. Pregnant or lactating females.
11. Not expected to survive within 48 hours of admission, or a presumed diagnosis of brain death.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse J Corry, MD, Principal Investigator — Allina Health
Locations (1):
- United Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annane D, Decaux G, Smith N; Conivaptan Study Group. Efficacy and safety of oral conivaptan, a vasopressin-receptor antagonist, evaluated in a randomized, controlled trial in patients with euvolemic or hypervolemic hyponatremia. Am J Med Sci. 2009 Jan;337(1):28-36. doi: 10.1097/MAJ.0b013e31817b8148. PMID 19057376
- [Background] Bulger EM, May S, Brasel KJ, Schreiber M, Kerby JD, Tisherman SA, Newgard C, Slutsky A, Coimbra R, Emerson S, Minei JP, Bardarson B, Kudenchuk P, Baker A, Christenson J, Idris A, Davis D, Fabian TC, Aufderheide TP, Callaway C, Williams C, Banek J, Vaillancourt C, van Heest R, Sopko G, Hata JS, Hoyt DB; ROC Investigators. Out-of-hospital hypertonic resuscitation following severe traumatic brain injury: a randomized controlled trial. JAMA. 2010 Oct 6;304(13):1455-64. doi: 10.1001/jama.2010.1405. PMID 20924011
- [Background] Chesnut RM, Temkin N, Carney N, Dikmen S, Rondina C, Videtta W, Petroni G, Lujan S, Pridgeon J, Barber J, Machamer J, Chaddock K, Celix JM, Cherner M, Hendrix T; Global Neurotrauma Research Group. A trial of intracranial-pressure monitoring in traumatic brain injury. N Engl J Med. 2012 Dec 27;367(26):2471-81. doi: 10.1056/NEJMoa1207363. Epub 2012 Dec 12. PMID 23234472
- [Background] Corry JJ, Varelas P, Abdelhak T, Morris S, Hawley M, Hawkins A, Jankowski M. Variable change in renal function by hypertonic saline. World J Crit Care Med. 2014 May 4;3(2):61-7. doi: 10.5492/wjccm.v3.i2.61. eCollection 2014 May 4. PMID 24892021
- [Background] Corry JJ. The use of targeted temperature management for elevated intracranial pressure. Curr Neurol Neurosci Rep. 2014 Jun;14(6):453. doi: 10.1007/s11910-014-0453-9. PMID 24740807
- [Background] Corry JJ. Use of hypothermia in the intensive care unit. World J Crit Care Med. 2012 Aug 4;1(4):106-22. doi: 10.5492/wjccm.v1.i4.106. eCollection 2012 Aug 4. PMID 24701408
- [Background] Costello-Boerrigter LC, Boerrigter G, Burnett JC Jr. Pharmacology of vasopressin antagonists. Heart Fail Rev. 2009 Jun;14(2):75-82. doi: 10.1007/s10741-008-9108-8. Epub 2008 Sep 3. PMID 18766438
- [Background] Adams Jr HP. Handbook of Cerebrovascular Disease. Ed.2 Marcel Dekker, Inc, New York, 2005
- [Background] Cumberland Pharmaceuticals, Inc. Vaprisol ® (conivaptan hydrochloride injection) [package insert]. Nashville, TN, April 2014.
- [Background] Dhar R, Murphy-Human T. A bolus of conivaptan lowers intracranial pressure in a patient with hyponatremia after traumatic brain injury. Neurocrit Care. 2011 Feb;14(1):97-102. doi: 10.1007/s12028-010-9366-x. PMID 20440600
- [Background] Diringer MN, Edwards DF. Admission to a neurologic/neurosurgical intensive care unit is associated with reduced mortality rate after intracerebral hemorrhage. Crit Care Med. 2001 Mar;29(3):635-40. doi: 10.1097/00003246-200103000-00031. PMID 11373434
- [Background] FDA. http://www.fda.gov/drugs/drugsafety/drugshortages/ucm050792.htm (2010)
- [Background] Fernandez N, Martinez MA, Garcia-Villalon AL, Monge L, Dieguez G. Cerebral vasoconstriction produced by vasopressin in conscious goats: role of vasopressin V(1) and V(2) receptors and nitric oxide. Br J Pharmacol. 2001 Apr;132(8):1837-44. doi: 10.1038/sj.bjp.0704034. PMID 11309256
- [Background] Galton C, Deem S, Yanez ND, Souter M, Chesnut R, Dagal A, Treggiari M. Open-label randomized trial of the safety and efficacy of a single dose conivaptan to raise serum sodium in patients with traumatic brain injury. Neurocrit Care. 2011 Jun;14(3):354-60. doi: 10.1007/s12028-011-9525-8. PMID 21409494
- [Background] Gazitua S, Scott JB, Chou CC, Haddy FJ. Effect of osmolarity on canine renal vascular resistance. Am J Physiol. 1969 Oct;217(4):1216-23. doi: 10.1152/ajplegacy.1969.217.4.1216. No abstract available. PMID 5824323
- [Background] Gebel JM Jr, Jauch EC, Brott TG, Khoury J, Sauerbeck L, Salisbury S, Spilker J, Tomsick TA, Duldner J, Broderick JP. Natural history of perihematomal edema in patients with hyperacute spontaneous intracerebral hemorrhage. Stroke. 2002 Nov;33(11):2631-5. doi: 10.1161/01.str.0000035284.12699.84. PMID 12411653
- [Background] Grande PO, Romner B. Osmotherapy in brain edema: a questionable therapy. J Neurosurg Anesthesiol. 2012 Oct;24(4):407-12. doi: 10.1097/01.ana.0000419730.29492.8b. PMID 22955195
- [Background] Hays A, Lazaridid C, et al. Osmotherapy in clinical practice: A survey of practitioners. Abstract Supplement. Volume 13. Neurocritical Care. 2010.
- [Background] Hemphill JC 3rd, Bonovich DC, Besmertis L, Manley GT, Johnston SC. The ICH score: a simple, reliable grading scale for intracerebral hemorrhage. Stroke. 2001 Apr;32(4):891-7. doi: 10.1161/01.str.32.4.891. PMID 11283388
- [Background] Kleindienst A, Fazzina G, Dunbar JG, Glisson R, Marmarou A. Protective effect of the V1a receptor antagonist SR49059 on brain edema formation following middle cerebral artery occlusion in the rat. Acta Neurochir Suppl. 2006;96:303-6. doi: 10.1007/3-211-30714-1_65. PMID 16671476
- [Background] Li YH, Sun SQ. [Expression of aquaporin - 4 protein in brain from rats with hemorrhagic edema]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2003 Sep;15(9):538-41. Chinese. PMID 12971848
- [Background] Liu X, Nakayama S, Amiry-Moghaddam M, Ottersen OP, Bhardwaj A. Arginine-vasopressin V1 but not V2 receptor antagonism modulates infarct volume, brain water content, and aquaporin-4 expression following experimental stroke. Neurocrit Care. 2010 Feb;12(1):124-31. doi: 10.1007/s12028-009-9277-x. PMID 19806476
- [Background] Marik PE, Rivera R. Therapeutic effect of conivaptan bolus dosing in hyponatremic neurosurgical patients. Pharmacotherapy. 2013 Jan;33(1):51-5. doi: 10.1002/phar.1169. PMID 23307545
- [Background] Mayer SA, Sacco RL, Shi T, Mohr JP. Neurologic deterioration in noncomatose patients with supratentorial intracerebral hemorrhage. Neurology. 1994 Aug;44(8):1379-84. doi: 10.1212/wnl.44.8.1379. PMID 8058133
- [Background] McGraw CP, Howard G. Effect of mannitol on increased intracranial pressure. Neurosurgery. 1983 Sep;13(3):269-71. doi: 10.1227/00006123-198309000-00009. PMID 6413884
- [Background] Migliati ER, Amiry-Moghaddam M, Froehner SC, Adams ME, Ottersen OP, Bhardwaj A. Na(+)-K (+)-2Cl (-) cotransport inhibitor attenuates cerebral edema following experimental stroke via the perivascular pool of aquaporin-4. Neurocrit Care. 2010 Aug;13(1):123-31. doi: 10.1007/s12028-010-9376-8. PMID 20458553
- [Background] Murphy T, Dhar R, Diringer M. Conivaptan bolus dosing for the correction of hyponatremia in the neurointensive care unit. Neurocrit Care. 2009;11(1):14-9. doi: 10.1007/s12028-008-9179-3. Epub 2009 Jan 4. PMID 19123060
- [Background] Naidech AM, Paparello J, Liebling SM, Bassin SL, Levasseur K, Alberts MJ, Bernstein RA, Muro K. Use of Conivaptan (Vaprisol) for hyponatremic neuro-ICU patients. Neurocrit Care. 2010 Aug;13(1):57-61. doi: 10.1007/s12028-010-9379-5. PMID 20568023
- [Background] Nathan BR. Cerebral correlates of hyponatremia. Neurocrit Care. 2007;6(1):72-8. doi: 10.1385/NCC:6:1:72. PMID 17356196
- [Background] National PBM Drug Monograph. Conivaptan Hydrochloride Injection (Vaprisol). 2006. [Appendix 6]
- [Background] Nau R, Desel H, Lassek C, Thiel A, Schinschke S, Rossing R, Kolenda H, Prange HW. Slow elimination of mannitol from human cerebrospinal fluid. Eur J Clin Pharmacol. 1997;53(3-4):271-4. doi: 10.1007/s002280050375. PMID 9476044
- [Background] Onuoho A, Human T, Dringer MN, Dhar R. Predictors of the Response to a Bolus of Conivaptan in Patients with Acute Hyponatremia. Abstract Supplement. Volume 13. Neurocritical Care. 2010.
- [Background] Rosenberg GA, Scremin O, Estrada E, Kyner WT. Arginine vasopressin V1-antagonist and atrial natriuretic peptide reduce hemorrhagic brain edema in rats. Stroke. 1992 Dec;23(12):1767-73; discussion 1773-4. doi: 10.1161/01.str.23.12.1767. Erratum In: Stroke 1993 Jun;24(6):913. PMID 1448828
- [Background] Ross WD. The right and the good. Hackett Pub Co Inc (July 1988). ISBN-13: 978-0872200586.
- [Background] Sheth KN, Kimberly WT, Elm JJ, Kent TA, Mandava P, Yoo AJ, Thomalla G, Campbell B, Donnan GA, Davis SM, Albers GW, Jacobson S, Simard JM, Stern BJ. Pilot study of intravenous glyburide in patients with a large ischemic stroke. Stroke. 2014 Jan;45(1):281-3. doi: 10.1161/STROKEAHA.113.003352. Epub 2013 Nov 5. PMID 24193798
- [Background] Strandvik GF. Hypertonic saline in critical care: a review of the literature and guidelines for use in hypotensive states and raised intracranial pressure. Anaesthesia. 2009 Sep;64(9):990-1003. doi: 10.1111/j.1365-2044.2009.05986.x. PMID 19686485
- [Background] Sun Z, Zhao Z, Zhao S, Sheng Y, Zhao Z, Gao C, Li J, Liu X. Recombinant hirudin treatment modulates aquaporin-4 and aquaporin-9 expression after intracerebral hemorrhage in vivo. Mol Biol Rep. 2009 May;36(5):1119-27. doi: 10.1007/s11033-008-9287-3. Epub 2008 Jun 24. PMID 18574711
- [Background] Szmydynger-Chodobska J, Chung I, Kozniewska E, Tran B, Harrington FJ, Duncan JA, Chodobski A. Increased expression of vasopressin v1a receptors after traumatic brain injury. J Neurotrauma. 2004 Aug;21(8):1090-102. doi: 10.1089/0897715041651033. PMID 15319008
- [Background] Taya K, Gulsen S, Okuno K, Prieto R, Marmarou CR, Marmarou A. Modulation of AQP4 expression by the selective V1a receptor antagonist, SR49059, decreases trauma-induced brain edema. Acta Neurochir Suppl. 2008;102:425-9. doi: 10.1007/978-3-211-85578-2_83. PMID 19388360
- [Background] Thiex R, Tsirka SE. Brain edema after intracerebral hemorrhage: mechanisms, treatment options, management strategies, and operative indications. Neurosurg Focus. 2007 May 15;22(5):E6. doi: 10.3171/foc.2007.22.5.7. PMID 17613237
- [Background] Taylor TN, Davis PH, Torner JC, Holmes J, Meyer JW, Jacobson MF. Lifetime cost of stroke in the United States. Stroke. 1996 Sep;27(9):1459-66. doi: 10.1161/01.str.27.9.1459. PMID 8784113
- [Background] Trabold R, Krieg S, Scholler K, Plesnila N. Role of vasopressin V(1a) and V2 receptors for the development of secondary brain damage after traumatic brain injury in mice. J Neurotrauma. 2008 Dec;25(12):1459-65. doi: 10.1089/neu.2008.0597. PMID 19118456
- [Background] Venkatasubramanian C, Mlynash M, Finley-Caulfield A, Eyngorn I, Kalimuthu R, Snider RW, Wijman CA. Natural history of perihematomal edema after intracerebral hemorrhage measured by serial magnetic resonance imaging. Stroke. 2011 Jan;42(1):73-80. doi: 10.1161/STROKEAHA.110.590646. Epub 2010 Dec 16. PMID 21164136
- [Background] Verbalis JG, Zeltser D, Smith N, Barve A, Andoh M. Assessment of the efficacy and safety of intravenous conivaptan in patients with euvolaemic hyponatraemia: subgroup analysis of a randomized, controlled study. Clin Endocrinol (Oxf). 2008 Jul;69(1):159-68. doi: 10.1111/j.1365-2265.2007.03149.x. Epub 2008 Jul 1. PMID 18034777
- [Background] Volbers B, Willfarth W, Kuramatsu JB, Struffert T, Dorfler A, Huttner HB, Schwab S, Staykov D. Impact of Perihemorrhagic Edema on Short-Term Outcome After Intracerebral Hemorrhage. Neurocrit Care. 2016 Jun;24(3):404-12. doi: 10.1007/s12028-015-0185-y. PMID 26381282
- [Background] Wilcox CS. Regulation of renal blood flow by plasma chloride. J Clin Invest. 1983 Mar;71(3):726-35. doi: 10.1172/jci110820. PMID 6826732
- [Background] Wright WL, Asbury WH, Gilmore JL, Samuels OB. Conivaptan for hyponatremia in the neurocritical care unit. Neurocrit Care. 2009;11(1):6-13. doi: 10.1007/s12028-008-9152-1. Epub 2008 Nov 12. PMID 19003543
- [Background] Yool AJ, Brown EA, Flynn GA. Roles for novel pharmacological blockers of aquaporins in the treatment of brain oedema and cancer. Clin Exp Pharmacol Physiol. 2010 Apr;37(4):403-9. doi: 10.1111/j.1440-1681.2009.05244.x. Epub 2009 Jun 29. PMID 19566827
- [Background] Zandor section of the Handbook of Experimental Pharmacology, Editors-in-chief: Starke, Klaus, Hofmann, Franz B. ISSN: 0171-2004.
- [Background] Zeltser D, Rosansky S, van Rensburg H, Verbalis JG, Smith N; Conivaptan Study Group. Assessment of the efficacy and safety of intravenous conivaptan in euvolemic and hypervolemic hyponatremia. Am J Nephrol. 2007;27(5):447-57. doi: 10.1159/000106456. Epub 2007 Jul 26. PMID 17664863
- [Background] Zeynalov E, Chen CH, Froehner SC, Adams ME, Ottersen OP, Amiry-Moghaddam M, Bhardwaj A. The perivascular pool of aquaporin-4 mediates the effect of osmotherapy in postischemic cerebral edema. Crit Care Med. 2008 Sep;36(9):2634-40. doi: 10.1097/CCM.0b013e3181847853. PMID 18679106
- [Derived] Corry JJ, Asaithambi G, Shaik AM, Lassig JP, Marino EH, Ho BM, Castle AL, Banerji N, Tipps ME. Conivaptan for the Reduction of Cerebral Edema in Intracerebral Hemorrhage: A Safety and Tolerability Study. Clin Drug Investig. 2020 May;40(5):503-509. doi: 10.1007/s40261-020-00911-9. PMID 32253717

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at a single medical institution between March 1, 2017 and November 7, 2018. The first participant was enrolled on March 22, 2017 and the last participant was enrolled on November 7, 2018.
Groups:
- Conivaptan Treatment Group: All seven patients in this arm will receive conivaptan as described in Interventions.
  Conivaptan: Patients will receive 20mg IV of the study drug every 12 hours equaling 40mg/day over 2 days (4 doses total), in addition to the standardized ICH management targets using the PI's version of standardized ICH management targets.Usual standard of care can include sedation and analgesia as needed, elevation of the head of the bed, mannitol and/or saline as needed to reduce ICP, and temperature control with antipyretics such as acetaminophen.
  The conivaptan bolus (20mg), which is premixed with 100ml of 5% dextrose in water, is infused (peripherally) over 30 minutes, most commonly through an already placed central line.
Period: Overall Study
Arm/Group | Conivaptan Treatment Group
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Conivaptan Treatment Group
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 58.5 [36 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Patient Tolerance of Conivaptan
Description: The number of participants with abnormal seizure activity and/or abnormal lab values and/or increase in infection rate and/or any drug-related adverse events.
Time Frame: Baseline to 168 hours post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Conivaptan Treatment Group
Number analyzed (Participants) | 7
Participants
  Abnormal Seizure Activity | 0
  Abnormal Lab Values | 0
  Infections | 1
  Drug-related Adverse Events | 0

2. Secondary Outcome: In-hospital Mortality
Description: All-cause deaths during hospitalization
Time Frame: Enrollment through hospital discharge, up to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Conivaptan Treatment Group
Number analyzed (Participants) | 7
Participants | 0

3. Secondary Outcome: Change in Cerebral Edema
Description: Changes in cerebral edema (CE) as measured on CT. Goal is a -5 to -10% change in CE over time. Change will be measured both as absolute change in volume, calculated as the final volume minus the baseline volume measure and converted to a percentage of the baseline volume measure.
Time Frame: Baseline to 168 hours post-enrollment
Measure: Mean (Full Range); unit: percentage of change from baseline
Arm/Group | Conivaptan Treatment Group
Number analyzed (Participants) | 7
percentage of change from baseline | -37.1 [-96.2 to 70.7]

4. Secondary Outcome: Cost
Description: Cost as measured by length of stay in the neuro ICU.
Time Frame: Enrollment through hospital discharge, up to 3 weeks
Measure: Mean (Full Range); unit: days
Arm/Group | Conivaptan Treatment Group
Number analyzed (Participants) | 7
days | 14.4 [9.7 to 28.9]

5. Secondary Outcome: Cost
Description: Cost as measured by:
  1. Need for external ventricular drain (EVD)/bolt or surgical procedures (craniectomy, clot evacuation,VPS) for reduction/management of CE.
  2. Need for central venous lines, arterial lines, peripherally inserted central venous catheter (PICC) lines, tracheostomy/percutaneous endoscopic gastrostomies (PEGs).
  3. Number of patients requiring a ventilator.
Time Frame: Baseline to 168 hours post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Conivaptan Treatment Group
Number analyzed (Participants) | 7
Participants
  EVD/bolt or surgical procedures | 0
  Lines or tracheostomy/PEG | 7
  Ventilator | 1

6. Secondary Outcome: Modified Rankin Scale (mRS) Score
Description: Modified Rankin Scale (0 to 6) at discharge from the hospital. A score of 0 indicates no disability and a score of 6 indicates the patient died. Functional independence is defined as a score of 2 or less.
Time Frame: At discharge from ICU and from hospital, up to 3 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Conivaptan Treatment Group
Number analyzed (Participants) | 7
score on a scale | 5 [3 to 5]

ADVERSE EVENTS:
Time Frame: Throughout study participation. For each patient this extended from enrollment to 3 months after enrollment.
Arm/Group | Conivaptan Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 7/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conivaptan Treatment Group (N=7)
Intracranial Hemorrhage Expansion (Nervous system disorders) | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2
Urinary Tract Infection (Infections and infestations) | 1
Catheterization, Central Venous (PICC) (Surgical and medical procedures) | 7 — Need for a peripherally inserted central catheter line
Tracheostomy (Surgical and medical procedures) | 3
Gastostomy (PEG) (Surgical and medical procedures) | 2
Increase in Cerebral Edema (Nervous system disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT03000283/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT03000283/SAP_001.pdf